CLINICAL TRIAL: NCT01709370
Title: Phase II Neoadjuvant Study of Letrozole in Combination With PD0332991 (Oral CDK 4/6 Inhibitor) for ER Positive, HER2 Negative Breast Cancer in Postmenopausal Women
Brief Title: Letrozole and CDK 4/6 Inhibitor for ER Positive, HER2 Negative Breast Cancer in Postmenopausal Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Organisation for Oncology and Translational Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OOTR-N007/LET-CDK
Record Dates: First submitted 2012-10-15; First posted 2012-10-18 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2012-10

CONDITIONS: ER Positive, HER2 Negative Breast Cancer
MeSH Terms: interventions — Letrozole; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Letrozole plus PD 0332991 (Experimental): Drug: Letrozole 2.5mg/d for 16 weeks before surgery plus PD 0332991 (CDK-4/6 inhibitor) 125 mg/d for 3 out of 4 weeks in repeated cycles for 16 weeks before surgery
  Interventions: Drug: Letrozole, PD 0332991

INTERVENTIONS:
Drug: Letrozole, PD 0332991

SUMMARY:
This is a phase II study evaluating the efficacy and safety of the pre-operative use of letrozole plus PD 0332991 (combination therapy)

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Primary tumor greater than 2 cm in diameter
* Histologically proven invasive breast cancer
* Positive estrogen receptor
* Negative HER-2 receptor
* ECOG performance status ≤ 1 or Karnofsky performance status ≥ 70%
* Laboratory values must be follows:

Absolute neutrophil count ≥ 1,500/mm3; Platelets ≥ 100,000/mm3; Hemoglobin ≥ 9 g/dL; Bilirubin ≤ 1.5 × institutional upper limit of normal (ULN); Serum Creatinine ≤ 1.5 × ULN; Alkaline phosphatase ≤ 2 × ULN; AST and ALT ≤ 2 × ULN; Normal finding of ECG - QTc ≤ 470 msec (based on the mean value of the triplicate ECGs); Left ventricular ejection fraction (LVEF) ≥ 60%.

* Able to give written informed consent form
* Able to follow prescription instructions reasonably well

Exclusion Criteria:

* Male
* Severe psychiatric disorder
* Prior history of other malignancy within 5 years of study entry, aside from basal cell carcinoma or the skin or carcinoma-in-situ of the uterine cervix
* Locally advanced breast cancer (T3N1 or Any T4 or Any N2, N3), or distant metastasis
* Multifocal or multicentric breast cancer except that the largest lesion is greater than 2cm
* Major surgery within 3 weeks of first study treatment
* Current use or anticipated need for:

Food or drugs that are known strong CYP3A4 inhibitors; drugs that are known strong CYP3A4 inducers

* Severe cardiovascular diseases in the previous 6 months
* Active inflammatory bowel disease or chronic diarrhea
* Renal Impairment
* Poor adrenal function
* Hepatitis B and/or hepatitis C carriers (unless with normal hepatic function)
* Known human immunodeficiency virus infection
* Known hypersensitivity to anti-aromatase drugs or any cell cycle inhibitor
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2012-02

PRIMARY OUTCOMES:
Objective response rates | Every 4 weeks before surgery

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Continuous during the study, up to 28 days after the last treatment

OTHER OUTCOMES:
Pathologic response rates | At time of definitive surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Unimed Medical Institute, Hong Kong, China